CLINICAL TRIAL: NCT02856971
Title: Rotating Hinge Knee Arthroplasty for Septic Revision After Total Knee Arthroplasty: a Retrospective Cohort About 50 Patients With 2 Years Follow up
Brief Title: Knee Hinge Prosthesis Following TKA Infection
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0522
Record Dates: First submitted 2016-08-02; First posted 2016-08-05 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-08

CONDITIONS: TKA Infection
Keywords: Hinge Knee Prosthesis; TKA infection; rotating hinge prosthesis; hinge knee arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Between 2009 and January 2016, the investigators included 49 patients from four hospitals in Lyon who had a Total Knee Arthroplasty (TKA) infection and who benefited of a knee arthroplasty revision with a rotating hinge prosthesis. This retrospective and descriptive cohort aims at studying the functional results after 2 years follow up.

ELIGIBILITY:
Inclusion Criteria:

- All the patients who had a rotating hinge knee arthroplasty for septic revision after total knee arthroplasty, proved by bacteriological samples or purulent drainage at involved site or other obvious clinical signs or radiological signs of infection

Exclusion Criteria:

- Patients who benefited of a hinge prosthesis following a unicompartmental prosthesis, following a mechanical issue on a total prosthesis

Ages: 45 Years to 91 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having a hinge knee prosthesis following an infection on a total knee prosthesis .
  Pre-operative characteristics studied :
  Clinical characteristics : medical and surgical history on the index knee included the strategy of the infection treatment (one step treatment vs two steps treatment)and general contributing factors of infection, frontal laxity, join motions, initial constraint of the infected TKA, skin condition ( skin necrosis, fistula, flap need, scar condition) paraclinical characteristics : bone defects, condition of knee extensor system ( continuance, height of patella, joint space height (when possible to measure)), prosthethic sealing or unsealing on CT-scan or scintigraphy, causal germ(s)
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2015-12; Primary Completion 2016-03 (Actual); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
functional results | at two years follow up
  Objective functional results : joint motions (Physician assessment)
functional results | at two years follow up
  Subjective functional results : satisfaction, patient expectations, functional activities. These items are based on the new IKS score

SECONDARY OUTCOMES:
infection control | after 2 years follow up
  presence or absence of clinical and/or biological signs of infection, recurrence of the infection or new secondary infection

CONTACTS AND LOCATIONS:
Overall Officials: Tristan Ferry, Pr, MD PhD, Principal Investigator — Hôpital de la Croix-Rousse
Locations (1):
- Centre de reference des infections ostéo-articulaires de Lyon,Groupement Hospitalier Nord - Hôpital de la Croix-Rousse - Bât. B, niveau 3 103 Grande-Rue de la Croix-Rousse, Lyon, France

REFERENCES:
- See also: Related Info — http://www.crioac-lyon.fr